CLINICAL TRIAL: NCT05379127
Title: "The (Cost-)Effectiveness of a Patient Empowered Protocol Without Routine X-rays for Follow-up of Adolescent Idiopathic Scoliosis Patients; A Pragmatic Randomized Trial"
Brief Title: Comparing Use of Radiographs Versus Patient Empowerment (CURVE)
Acronym: CURVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Trialbureau Zorgevaluatie Nederland (Unknown); Nederlandse Orthopaedische Vereniging (Unknown); Vereniging Scoliose Patiënten (Unknown); Dutch Adolescent Idiopathic Scoliosis (AIS) Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 80-87600-98-19048
Record Dates: First submitted 2022-05-06; First posted 2022-05-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Spine; Quality of Health Care; Cost-Benefit Analysis; Patient Participation; Radiology
MeSH Terms: conditions — Scoliosis; Patient Participation

STUDY DESIGN:
Intervention Model Description: A multicentre pragmatic randomized trial design with two arms, combined with a patient preference cohort for each arm (partially randomized preference trial; PRPT).
  The PRPT consists of three separate randomized controlled trials (RCTs) including patients in the pre-treatment phase, post-brace phase or post-operative phase. Alongside the RCTs prospective preference cohorts are included for each treatment arm (patient empowered follow up [PE-FU] or standard follow up [standard FU]). In the preference cohorts all patients are monitored who are not willing (i.e. who have a preference for either the standard FU or PE-FU) to be randomized to either treatment arm, but who are still willing to participate in the study. By including preference cohorts the generalizability of study results is studied while the internal validity is assured.
  * Half of participants (n=406) allocation: randomized (RCT)
  * Half of participants (n=406) allocation: based on preference (preference cohorts)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard follow-up (Other): standard care during follow-up
  Interventions: Other: Standard follow-up
- Patient-empowered follow-up (Experimental)
  Interventions: Other: Patient-empowered follow up

INTERVENTIONS:
Other: Patient-empowered follow up — The patient-empowered follow-up protocol consists of patient-reported outcome measures (PROMs), self-assessment tools and clinical assessment including physical examination. Radiographs will only be taken when progression of the scoliosis (curve progression) or postoperative complications are suspected based on test results and based on the criteria of so called 'sense of alarm'.
  Note: Sense of alarm ('niet pluis') is based on any deterioration on the above-mentioned PROMs, self-assessment tool, and clinician-based measurement instruments, which is a signal for the treating physician to consider when a radiograph is appropriate. Sense of alarm is described as any other concern by the orthopaedic surgeon, parent or child which warrants a radiograph. For both the Bunnell Scoliometer (clinical assessment tool) and the Scolioscoop (patient self-assessment tool) a threshold of ≥4° is used.
  Arms: Patient-empowered follow-up
Other: Standard follow-up — Routine radiographs are taken at each follow up visit during standard care (to detect possible curve progression or rule out postoperative complications).
  Arms: Standard follow-up

SUMMARY:
Objective: To evaluate the (cost-)effectiveness of a new patient-empowered follow up (FU) protocol in patients with Adolescent idiopathic Scoliosis (AIS) that is based on patient-reported outcome measures (PROMs), self-assessment tools and physical examination, which is compared to standard FU care by: 1) Effect evaluation, 2) Economic evaluation, 3) Implementation (process) evaluation.

Study design: A multicentre pragmatic randomized trial design with two arms, combined with a patient preference cohort for each arm (partially randomized preference trial [PRPT]).

Study population: A total of 812 AIS patients (age 10-18 years) treated by the Dutch AIS Consortium, representing the scoliosis treatment centres in the Netherlands, will be included.

Three subgroups of AIS patients are distinguished, which are monitored over two years:

1. Pre-treatment group: adolescents with curve 10-25° (n=132 per arm; total n=264)
2. Post-brace treatment group (n=122 per arm; total n=244)
3. Post-surgery group (n=152 per arm; total n=304)

Intervention: The new patient-empowered FU protocol (PE-FU) is based on PROMs, self-assessment tools and clinical assessment including physical examination. The protocol aims to detect curve progression or postoperative complications based on these patient-based and clinical parameters to substitute the need to obtain routine x-rays. X-rays will only be taken when progression or postoperative complications are suspected in the pre- and post-intervention groups based on predefined criteria. The standard FU protocol consists of routine full-spine radiographs and routine clinical evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adolescent idiopathic scoliosis (AIS).
* Age: 10-18 years old.
* Patients scheduled for follow up in one of the participating centres.
* Understanding of the Dutch language.
* Signed informed consent.
* Biplanar (Posterior-Anterior [PA] and Lateral) full-spine x-rays within the last 3 months.

Specifically for the pre-treatment group:

* Girls aged ≤14 years (i.e. 10-14 years) and boys <16 years (i.e. 10-15 years). These patients still have generally 2 years of remaining skeletal growth. Patients above this age with a curve below 25 degrees have a limited risk for progression
* Girls: pre-menarche up to 6 months post-menarche (to estimate end of growth)
* A primary coronal curve of 10-25 degree.

Specifically for the post-brace group:

* Patients aged 12-18 years
* Within 3 months after termination of brace treatment
* Minimum of 6 months of brace treatment

Specifically for the post-surgery group:

• Patients aged 12-18 years

Exclusion Criteria:

* Patients with juvenile or infantile idiopathic scoliosis with the diagnosis of onset under the age of 10.
* Patients who are undergoing brace treatment. These patients are not included because of the need to monitor brace therapy with radiographs.
* Patients who have undergone previous spinal surgery and are undergoing revision surgery.
* Skeletally mature patients.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 812 (Estimated)
Dates: Start 2022-07-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of radiographs that has led to treatment consequences | 24 months
  the proportion will serve as an indication of the sensitivity of the new PE-FU protocol and standard FU protocol. The number of x-rays that has led to treatment will be divided by the total number of x-rays in each subgroup to calculate the primary outcome.

SECONDARY OUTCOMES:
The safety of the standard and the new protocol | for pre-treatment and the post-brace group at 6, 12,18 and 24 months and for the postsurgery group at 3,12 and 24 months
  The number of false negative radiological findings with treatment consequences not detected by any of the protocols at the end of the study period. This consists of the proportion of patients with delayed detection of progression or post-operative complications (e.g. a pseudo-arthrosis, curve progression, adding on), which requires treatment or increased vigilance.
The specificity, negative predictive value and positive predictive value of the standard and new patient empowered follow up protocol. | 24 months
The change in readiation exposure | 24 months
  The exposure in the new follow up will be compared to standard care using reference values
Participants perspective: Numeric pain rating scale [NPRS 0-10] | 24 Months
  Numeric rating scale for back pain, score range 0-10, 0 no pain at all and 10 wrost pain imaginable.
Participants perspective: condition-specific quality of life [SRS-22r] | 24 months
  Scoliosis Research Society 22 items about function, pain, self image, mental health and statifaction.
Participants perspective: health-related quality of life [EQ5D-5L] | 24 months
  Dutch EQ-5D-5L using the Dutch utility score.
Participants perspective: Scoliosis Appearance questionnaire short version [short SAQ]) | 24 months
  Dutch version of the scoliosis appearance questionnaire.
Global perceirved effect [GPE] | 24 months
  the recovery and statisfaction of the participant during and after treatment.
educational status | 24 months
  questions related to absence from school, absence from physical education classes, frequency of missing school exams, necessity to repeat a class, support and alternatives provided by the school, and return to school and sport after surgery.
Self-assessment tool: Scolioscoop | or pre-treatment and the post-brace group at 6, 12,18 and 24 months and for the postsurgery group at 3,12 and 24 months
  Change in the trunk asymmetry (degrees).
Cost-Benefit analysis: Patient outcome analysis using Quality-Adjusted Life Years (QALY). | 24 months
  Patient outcome analysis is based on EQ5D-5L.
Cost-Benefit analysis: Cost analysis | 24 months
  The costs will be assessed from a societal and a healthcare perspective. From the societal perspective, intervention, other healthcare, unpaid productivity, informal care, and absenteeism costs will be included, whereas only costs accruing to the formal Dutch healthcare sector will be included for the healthcare perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Miranda L van Hooff, PhD, Principal Investigator — Radboud University Medical Center; Marinus de Kleuver, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (23):
- Netherlands (23):
  - Isala, Zwolle, Drenthe
  - Flevo ziekenhuis, Almere Stad, Flevoland
  - Rijnstate, Arnhem, Gelderland
  - St Jansdal, Harderwijk, Gelderland
  - Maastricht UMC+, Maastricht, Limburg
  - Viecuri, Venlo, Limburg
  - Sint Maartenskliniek, Boxmeer, North Brabant
  - Amphia, Breda, North Brabant
  - ETZ Elisabeth, Tilburg, North Brabant
  - Noordwestziekenhuis groep, Alkmaar, North Holland
  - OLVG, Amsterdam, North Holland
  - Amsterdam UMC, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Dijklander, Hoorn, North Holland
  - Albert Schweitzer ziekenhuis, Dordrecht, South Holland
  - Groene Hart ziekenhuis, Gouda, South Holland
  - Leiden UMC, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Maasstad ziekenhuis, Rotterdam, South Holland
  - Juliana kinderziekenhuis, The Hague, South Holland
  - Meander, Amersfoort, Utrecht
  - UMC Groningen, Groningen
  - UMC Utrecht, Utrecht